CLINICAL TRIAL: NCT03706105
Title: Integrating Stroke Survivors Into Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Novant Health Heart and Vascular Institute (Unknown); American Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Elizabeth Regan, Physical Therapist, PhD Candidate, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1001
Record Dates: First submitted 2018-04-25; First posted 2018-10-15 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - Cardiac Rehabilitation (Experimental)
  Interventions: Behavioral: Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — 3 x week ~1 hour of exercise + education

SUMMARY:
The intervention trial will examine the effectiveness and feasibility of integrating stroke survivors into an existing hospital-based cardiac rehabilitation program at Novant Health in Charlotte, NC. Stroke survivors will be recruited through hospital system providers and physical therapists (PTs) for entry into a multidisciplinary, three-month cardiac rehabilitation program. This program consists of three sessions per week of supervised cardiovascular endurance and strength training, stretching, relaxation and education. Participants will be stroke survivors, have completed formal physical and occupational rehabilitation (if applicable), and have treating provider approval.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* Completion of physical and occupational therapy (if applicable)
* Clearance by treating medical provider
* Ability to walk at least 40 meters independently (with or without assistive device)
* Ability to transfer sit to stand without assistance
* Ability to follow instructions and provide information on exertion, pain and distress

Exclusion Criteria:

* Acute medical problem rendering exercise unsafe
* Significant pain that prevents standing or interferes with movement
* History of additional, non-stroke, neurological condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
6-minute walk Test | Change in 6-minute walk test at 3 months
  Aerobic and Walking Capacity Measure

SECONDARY OUTCOMES:
Walking Speed | Change in Walking Speed at 3 months
  Self-Selected walking speed for 10 meters
Timed Up and Go | Change in timed up and go at 3 months
  Mobility Measure: timed movement from seated in a chair, walk 10 feet and return to sitting in a chair.
Stroke Impact Scale | Change in Stroke Impact Scale at 3 months
  Quality of Life Questionnaire evaluating difficulty after stroke in 8 domains: strength, hand function, activities of daily living, mobility, communication, emotion, memory/thinking, participation/role function. Score is 0-100 in each domain and is transformed using the equation Domain score = (mean item score - 1)/4 * 100. Higher Scores indicate less impact of stroke.
Fatigue Severity Scale | Change in Fatigue Severity Scale at 3 months
  A scale measuring the perceived impact of fatigue on life activities. Total score is 9-63 with a higher score indicating more fatigue severity and impact.
Activities Specific Balance Confidence (ABC) Scale | Change in ABC Scale at 3 months
  The Activities Specific Balance Confidence scale measures an individual's confidence in performing 16 activities without loss of balance. Possible scores are 0-100 with higher scores indicating higher balance confidence.
Readiness for Change Questionnaire | Change in Readiness/Confidence in Behaviors at 3 months
  The readiness for change questionnaire evaluates self-perception of readiness and confidence in exercise, physical activity and overall wellness behaviors. Readiness score is 3-15 with higher scores indicating higher readiness, and confidence score 3-9 with a higher score indicating more confidence in behavior.
Patient Health Questionnaire 9 (PHQ9) | Change in PHQ9 at 3 months
  The patient health questionnaire is a 9 question self report measure of depression and depression severity. The score is 0-27 with a higher score indicating more severe depression.
Ferrans and Powers Quality of Life Questionnaire | Change in Ferrans and Powers Quality of Life Questionnaire at 3 months
  Ferrans and Powers Quality of Life questionnaire is a measure of satisfaction and importance of 7 domains (health, healthcare, self-care, energy, family/friends support, engagement in life activities, happiness). Raw scores are converted to overall scores by weighting satisfaction by importance and adjusting for unanswered questions. Total scores are 0-30 with higher scores indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy L Fritz, PT, PhD, Study Director — University of South Carolina; Elizabeth Regan, DPT, Principal Investigator — University of South Carolina
Locations (1):
- Novant Health Heart and Vascular Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Regan EW, Handlery R, Stewart JC, Pearson JL, Wilcox S, Fritz S. Integrating Survivors of Stroke Into Exercise-Based Cardiac Rehabilitation Improves Endurance and Functional Strength. J Am Heart Assoc. 2021 Feb 2;10(3):e017907. doi: 10.1161/JAHA.120.017907. Epub 2021 Jan 27. PMID 33499647